CLINICAL TRIAL: NCT02412813
Title: A Prospective, Randomized, Multi-Center, Metal Hypersensitivity Study Comparing OXINIUM and Cobalt Chrome Femoral Components in Failed Total Knee Arthroplasty
Brief Title: LEGION™ Revision Metal Hypersensitivity Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Overhaul of Study Design
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-4050-05
Record Dates: First submitted 2015-03-05; First posted 2015-04-09 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-03

CONDITIONS: Total Knee Replacement Revision
Keywords: hypersensitivity; metal sensitivity; arthroplasty; implant-related hypersensitivity; metal-on-metal implants; knee revision
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LEGION OXINIUM femoral component (Active Comparator)
  Interventions: Device: LEGION OXINIUM
- LEGION Cobalt Chrome femoral components (Active Comparator)
  Interventions: Device: LEGION Cobalt Chrome

INTERVENTIONS:
Device: LEGION OXINIUM — Investigational Group
  Arms: LEGION OXINIUM femoral component
Device: LEGION Cobalt Chrome — Control Group
  Arms: LEGION Cobalt Chrome femoral components

SUMMARY:
This is a prospective, randomized, multi-center, metal hypersensitivity study comparing OXINIUM and cobalt chrome femoral components in subjects with failed total knee arthroplasty (TKA).

DETAILED DESCRIPTION:
A total of 230 subjects will be randomized (1:1) to receive either an OXINIUM or cobalt chrome femoral components as part of their LEGION revision procedure. The objective of this study is to assess a lower serum metal ion concentration level in at least one of the three major mLTTs (Co, Cr or Ni) over 5 years in subjects receiving OXINIUM versus Cobalt Chrome femoral components as part of the LEGION Revision Total Knee System.

ELIGIBILITY:
Inclusion Criteria:

* Subject is skeletally mature
* Subject is willing to sign and date an IRB/EC approved consent form
* Subject is a candidate for a revision knee replacement
* Subject has met an acceptable preoperative medical clearance and is free or treated for cardiac, pulmonary, hematological, infection, or other conditions that would pose excessive operative risk
* Subject agrees to adhere to the 10-year study visit schedule

Exclusion Criteria:

* Subject with a known metal hypersensitivity
* Subject requires a known bilateral revision TKA
* Subject has severe pronation of the ipsilateral foot or any other relevant clinical condition contributing to abnormal ambulation
* Subject has active infection or sepsis (treated or untreated)
* Subject with an immunosuppressive disorder
* Subject has presence of malignant tumor, metastatic, or neoplastic disease
* Subject has conditions that may interfere with the TKA survival or outcome (i.e., Paget's or Charcot's disease, vascular insufficiency, muscular atrophy, uncontrolled diabetes, moderate to severe renal insufficiency or neuromuscular disease)
* Subject has had intra-articular corticosteroid therapy (or any other intra-articular therapy) in the study knee within 3 months of study enrollment
* Subject has inadequate bone stock to support the device and would require significant augmentation to correct the joint Female subject is of child-bearing age and unwilling to use an approved method of contraception
* Subject has an emotional or neurological condition that would pre-empt their ability or willingness to comply with the study
* Subject is severely overweight (BMI>40)
* Subject is currently enrolled in another investigational drug, biologic, or device study or has been treated with an investigational product in the past 30 days
* Subject is facing current or impending incarceration

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Major modified Lymphocyte Transformation Tests (Cobalt, Chromium and Nickel) measurements | 3,650 Days
  Metal hypersensitivity will be concluded if at least one of these three measurements is statistically significant

SECONDARY OUTCOMES:
Minor modified Lymphocyte Transformation Tests (Aluminum, Iron, Molybdenum, Vanadium and Zirconium) | 3,650 Days
  changes in mean mLTTs serum concentration values from baseline to each subsequent assessment
Changes in mean serum bio-markers from baseline to each subsequent assessment | 3,650 Days
Skin lesion evaluation to measure hypersensitivity | 3,650 Days
Revision of LEGION Revision Knee System for any reason at each post-surgical assessment | 3,650 Days
Improves in mean 2011 Knee Society Score (2011 KSS) from baseline to each subsequent assessment | 3,650 Days
Anteroposterior, lateral and skyline knee views are assessed by radiographs | 3,650 Days
All adverse event reporting from surgery to 10 year post-surgery | 3,650 Days

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Turgeon, MD, Principal Investigator — Orthopaedic Innovation Centre
Locations (3):
- United States (2):
  - Rothman Institute, Egg Harbor, New Jersey
  - Columbia University Medical Center, New York, New York
- Orthopaedic Innovation Centre, Winnipeg, Manitoba, Canada